CLINICAL TRIAL: NCT02806674
Title: A Relevance Study Between the Result of Clinical Drug Intervention and Next-generation Sequencing Technology Focused on Refractory Helicobacter Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Collaborators: People Hospital of Luohu,Shenzhen (Unknown); Shenzhen Second People's Hospital (Other); Longhua Branch of Shenzhen People Hospital (Unknown); The People Hospital of Baoan Shenzhen (Other); Zhiyuan Medical Inspection Institute (Other)
Responsible Party: Principal Investigator, TaoLYU, Deputy Director of the Department of Gastroenterology, The University of Hong Kong-Shenzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHongKongShenzhen
Record Dates: First submitted 2016-06-09; First posted 2016-06-21 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Gastritis
Keywords: Helicobacter pylori; Antibiotic resistance; Sequencing
MeSH Terms: conditions — Gastritis

ARMS (2):
- Successful treatment (Experimental)
  Interventions: Device: The eradication times of the patients; Device: The result of 13C-urea breath test after treatment
- Refractory infection of H.pylori (Experimental)
  Interventions: Device: The eradication times of the patients; Device: The result of 13C-urea breath test after treatment

INTERVENTIONS:
Device: The eradication times of the patients — The patients who have failed more than 2 eradication courses with standardized treatment were the refractory infection of H. pylori group,and patients who succeeded at the first standardized treatment were the successful treatment group
Device: The result of 13C-urea breath test after treatment — The intervention focused on the results from the result of 13C-urea breath test after treatment.The two groups were treatment based on the antibiotic susceptibility testing. Eight weeks after treatment,a 13C-urea breath test was performed on patients.The successful treatment group were patients with negative in 13C-urea breath tests in the first treatment. The refractory infection of H. pylori group were treatment failure patients after the second standardized treatment.

SUMMARY:
Approximately 50% of people in the world are infected with H. pylori, and its eradication rate fail to exceed 80% and even fails into an unacceptable range.Various risk factors for infection include lower socioeconomic status, younger age, and geographic location.In the present study, investigators aimed to perform a prevalence survey about risk factors for H. pylori infection.To obtain the higher eradication of H. pylori and find out the relevance between the diverse infection and clinical drug focused on refractory H. pylori infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~70 years old, male or female, untreated patients.
2. Symptoms of abdominal pain, bloating, acid reflux,belching,nausea,vomiting,heartburn, chest pain, vomiting, melena, etc.
3. Unused antibiotics, bismuth, H2 receptor antagonists or PPI by nearly 4 weeks
4. 13C-labelled urea breath test positive.
5. Agreed to Helicobacter pylori culture and sensitivity testing taken by endoscopy gastric biopsy specimens,and the result of culture was positive.
6. Agreed to Helicobacter pylori eradication therapy and cooperate with the eradication efficacy follow-up survey.

Exclusion Criteria:

1. Severe heart, liver, kidney dysfunction.
2. Pregnant or lactating women.
3. Complications of bleeding, perforation, pyloric obstruction, cancer.
4. Esophageal,gastrointestinal surgery history.
5. Patients can not properly express their complaints,such as psychosis, severe neurosis.
6. Taking NSIAD or alcohol abusers.
7. Allergic to penicillin or either drugs of the 6 antibiotic tested by susceptibility testing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1845 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The eradication rate of H. pylori reach to 95% | 1.5 year
  The eradication rate of untreated cases reach to 98%.The eradication rate of refractory cases reach to 90%.
Obtain the first resistant pattern to antibiotics in shenzhen area | 1.5 year
  The results of antibiotic susceptibility testing were analyzed in this study.More than 1800 patients were participated,these patients were representative in five hospitals of shenzhen area.
The proportion of mix infection of H pylori in a total of 40 patients in two groups | 2.5 year
  Analyzed the next-generation sequencing data,obtain the proportion of mixed infection with different H. pylori strain in refractory cases.

SECONDARY OUTCOMES:
The incidence of adverse effects in the eradicate treatment | 2.5 year
  A telephone interview was conducted at 4 weeks after treatment.And the 1845 patients was investigated using questionnaires of symptom checklist.A statistics table will be got.
The difference between microbial genes of different patients | 3 year
  By 2 or 3 metabolic pathways with significant differences, selected 40-50 different genes.
The relevance between mixed infection, microflora structure and risk factors | 3 year
  Analyzed the next-generation sequencing data,obtain the results of mixed infection and microflora structure in a total of 40 patients in two groups.And the patients was investigated using questionnaires of risk checklist.The collected data were subsequently analyzed using SPSS. For checking the relationship between mixed infection, microflora structure and risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Lyu, Doctor, Principal Investigator — The University of HongKong-Shenzhen Hospital
Locations (4):
- China (4):
  - The People Hospital of Baoan Shenzhen, Shenzhen, Guangdong
  - Longhua Branch of Shenzhen People Hospital, Shenzhen, Guangdong
  - People Hospital of Luohu,Shenzhen, Shenzhen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong